CLINICAL TRIAL: NCT00221676
Title: Effectiveness of Influenza Vaccination (Alfarix)in Preventing Clinical Influenza Cases Among General Practitioners: Non-Randomized Clinical Trial.
Brief Title: Effectiveness of Influenza Vaccination Among General Practitioners
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other); Eurogenerics NV (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHA-UA-20011207
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2006-11-28 (Estimated); Status verified 2005-09

CONDITIONS: Influenza
Keywords: influenza vaccine; general practitioner
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: Alfarix

SUMMARY:
Besides the personal protection, influenza vaccination especially needs to prevent transmission of influenza between GPs and their patients. The question remains if the vaccine is adding substantial benefit to the natural acquired immunity of GPs. Doubts are raised if an inactivated vaccine, which elicit especially humoral immune response, can give enough protection against virus replication and subclinical influenza infections. Until now no effectiveness studies of influenza vaccination were performed among GPs. This study will assess the effectiveness of an inactivated influenza vaccine in GPs against clinical respiratory tract infections and more particular against influenza cases with influenza positive nose and throat swabs (diagnosed by RT-PCR).

DETAILED DESCRIPTION:
Two important aspects emerge when considering influenza vaccination of general practitioners as advocated by many guidelines. Besides the personal protection the vaccine especially needs to prevent transmission of influenza between GPs and their patients. In long-term elderly hospitals a possible benefit of influenza vaccination of the healthcare workers was noticed in reducing mortality among the elderly. But this specific situation is not fully transmissible to the general practice.

GPs, having yearly close contact with several influenza cases, built up a high basic immunity and probably only suffer from minor symptoms. The question remains if the vaccine is adding substantial benefit to this natural acquired immunity. In addition doubts are raised in the literature if an inactivated vaccine, which elicit especially humoral immune response, can give enough protection against virus replication and subclinical influenza infections. Until now no effectiveness studies of influenza vaccination were performed among GPs. High time to look more closer to these issues.

Comparisons: the effectiveness of an inactivated influenza vaccine compared with no vaccine in GPs against clinical respiratory tract infections and more particular against influenza cases with influenza positive nose and throat swabs (diagnosed by RT-PCR), besides serological defined influenza cases and taking important independent variables into account

ELIGIBILITY:
Inclusion Criteria:general practitioner with an active practice in Flanders, Belgium -

Exclusion Criteria:other specialists in medicine

-

Ages: 25 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2002-07; Study Completion 2004-06

PRIMARY OUTCOMES:
number of respiratory tract infections
number of influenza cases defined as a RTI with positive nose and throat swabs
number of influenza cases defined as a RTI with 4-fold IgG titre rise

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Michiels, Dr., Principal Investigator — University of Antwerp, Department of family medicine

REFERENCES:
- [Result] Michiels B, Philips H, Coenen S, Yane F, Steinhauser T, Stuyck S, Denekens J, Van Royen P. The effect of giving influenza vaccination to general practitioners: a controlled trial [NCT00221676]. BMC Med. 2006 Jul 10;4:17. doi: 10.1186/1741-7015-4-17. PMID 16831228